CLINICAL TRIAL: NCT02247830
Title: Prophylactic Interventions in the Management of Radiodermatitis in Patients With Breast or Head and Neck Cancer: a Randomized Clinical Trial
Brief Title: Management Radiodermatitis in Patients With Breast or Head and Neck Cancer
Acronym: PRBHNC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Elaine Barros Ferreira, Nurse, University of Brasilia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: radiodermatite01
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Radiodermatitis
Keywords: Radiodermatitis; Head and neck neoplasms; Radiotherapy; Urea; Matricaria; Breast Neoplasms; chamomilla; chamomile
MeSH Terms: conditions — Radiodermatitis; Head and Neck Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Chamomilla recutita gel (Experimental): Experimental Group 01: usual care + topical application of the gel recutita chamomile. Such intervention will be characterized by topical application of the gel C. recutita, concomitantly to the initiation of radiotherapy, should be applied on the irradiated three times daily throughout the period of realization of radiotherapy sessions area, and nursing consultations with equipment instructional (usual care).
  Interventions: Other: Chamomilla recutita gel
- 2 Urea cream (Experimental): Experimental Group 02: usual care + Topical Application of Urea cream. The intervention will be characterized by topical application of urea-based cream on the area irradiated three times daily throughout the period of realization of radiotherapy sessions, in addition to nursing consultation with instructional material (usual care).
  Interventions: Drug: Urea cream
- Control Group (Usual Care) (No Intervention): The usual care consists of nursing consultation with instructional material (Manual guidelines) that is already done systematically in service. This query is made with all patients starting radiotherapy. Here, guidelines are provided about skin care and hydration, using topical moisturizing soap solution over the bath. Such information is contained in the manual that is provided to the patient during the consultation.

INTERVENTIONS:
Other: Chamomilla recutita gel — Such intervention will be characterized by topical application of C. recutita gel, concomitantly to the initiation of radiotherapy, should be applied on the irradiated region three times daily throughout the period of realization of radiotherapy sessions area, and nursing consultations with equipment instructional (usual care).
  Other Names: matricaria gel; chamomilla gel; chamomile gel
  Arms: 1 Chamomilla recutita gel
Drug: Urea cream — Experimental Group 02: usual care + Topical Application of Urea cream. The intervention will be characterized by topical application of urea-based cream on the irradiated region three times daily throughout the period of realization of radiotherapy sessions, in addition to nursing consultation with instructional material (usual care).
  Other Names: Urea cream based
  Arms: 2 Urea cream

SUMMARY:
It aims to evaluate the efficacy of the chamomile recutita gel and urea cream in the prevention of radiodermatitis in patients with breast cancer or head and neck cancer undergoing radiotherapy.

Prophylactic Trial will consist of a control group and two experimental groups, namely control group (usual care), Experimental Group 01 (usual care + topical application of the gel C. recutita) and Experimental Group 02 (usual care + topical application of Urea based cream).

The doses used in the different compounds are being in test since february 2014 by a dose-response curve study, using 6 groups with three doses of urea cream and three doses of C. recutita gel.

The study will be conducted at the Center for High Complexity Oncology at University Hospital of Brasília (CACON/HUB), Brazil. The degree of radiodermatitis is evaluated weekly, according to established criteria to classify the effects of radiotherapy, which identifies grades 0, 1, 2 , 3 and 4, according to the score of the Radiation Therapy Oncology Group - RTOG. To evaluate the skin reaction will also be applied scale Common Terminology Criteria for Adverse Events (CTCAE) and Radiation-Induced Skin Reaction Assessment Scale (RISRAS).

DETAILED DESCRIPTION:
It is considered that patients undergoing radiotherapy in use gel based on C. recutita or use of cream based urea three times a day, concomitant radiotherapy, would present the following hypotheses:

* Null: equal incidence and severity of radiodermatitis when compared to the control group (usual care);
* Alternative 1: low incidence and severity of radiodermatitis when compared to patients who comprised the control group (usual care).
* Alternative 2: lower incidence and severity of radiodermatitis between the experimental groups (urea and chamomile).

ELIGIBILITY:
Inclusion Criteria:

* Being an adult, over the age of 18 years old;
* Owning diagnosis of malignant breast or head and neck;
* Being first referred to the radiotherapy protocol;
* Agree to participate, expressing his acceptance by signing the Informed Consent Form (ICF);
* Present absence of dermatitis to initiation of radiotherapy;
* Demonstrate understanding of and conditions to continue the intervention in their home environment when needed.

Exclusion Criteria:

* Reports of previous hypersensitivity reaction or presentation, during the research, adverse reaction to chamomile or any plant of the Asteraceae or compositae family, or urea;
* Medical prescription for the procedure of data collection, some kind of intervention to prevent radiodermatitis;
* Withdrawal of the patient to remain in the study, independent of time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of radiodermatitis | 5 weeks
  Time of occurrence of radiodermatitis second dose of radiation (or its absence during radiotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Barros Ferreira, RN, Principal Investigator — University of Brasilia; Paula Elaine Diniz dos Reis, RN, PhD, Study Director — University of Brasilia; Marcia A Ciol, PhD, Study Director — University of Washington
Locations (1):
- University Hospital of Brasília, Brasília, Brazil